CLINICAL TRIAL: NCT00544596
Title: A Phase 1 Study of R-(-)-Gossypol (AT-101) in Combination With Cisplatin and Etoposide in Patients With Advanced Solid Tumors and Extensive-Stage Small Cell Lung Cancer
Brief Title: R-(-)-Gossypol Acetic Acid, Cisplatin, and Etoposide in Treating Patients With Advanced Solid Tumors or Extensive Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00273; NCI-2009-00273 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CO07901; 2007-0145; CDR0000570006; CO 07901 (Other: University of Wisconsin Hospital and Clinics); 8062 (Other: CTEP); P30CA014520 (NIH); U01CA062491 (NIH)
Record Dates: First submitted 2007-10-13; First posted 2007-10-16 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2012-06

CONDITIONS: Extensive Stage Small Cell Lung Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — gossypol acetic acid; Cisplatin; Etoposide

ARMS (1):
- Treatment (R-(-)-gossypol acetic acid, cisplatin, etoposide) (Experimental): Patients receive oral R-(-)-gossypol twice daily on days 1-3, cisplatin IV over 60 minutes on day 1*, and etoposide IV over 30 minutes on days 1*-3. Treatment repeats every 21 days for up to 6 courses during the dose escalation and 4 courses in the expanded extensive stage small cell lung cancer cohort, in the absence of disease progression or unacceptable toxicity.
  Blood samples are collected on day 1 of courses 1 and 2 for pharmacokinetic analysis, biomarker assays, and correlative studies.
  After completion of study treatment, patients are followed for 30 days.
  [Note: *Cisplatin and etoposide will be started on day 2 during course 1; they will be given on day 1 during all subsequent courses.]
  Interventions: Drug: R-(-)-gossypol acetic acid; Drug: cisplatin; Drug: etoposide

INTERVENTIONS:
Drug: R-(-)-gossypol acetic acid — Given orally
  Other Names: AT-101
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213

SUMMARY:
This phase I trial is studying the side effects and best dose of R-(-)-gossypol acetic acid when given together with cisplatin and etoposide in treating patients with advanced solid tumors or extensive stage small cell lung cancer. R-(-)-gossypol acetic acid may stop the growth of cancer by blocking blood flow to the tumor. Drugs used in chemotherapy, such as cisplatin and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving R-(-)-gossypol acetic acid together with combination chemotherapy may help kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) or recommended phase II dose (RP2D) of AT-101 (R-(-)-gossypol) when combined with cisplatin and etoposide in patients with advanced, refractory solid tumors and/or extensive stage small cell lung cancer (ES-SCLC). In addition, to determine the MTD or RP2D of AT-101 when combined with cisplatin, etoposide, and Neulasta.

II. To evaluate the toxicity and tolerability of AT-101 in combination with cisplatin and etoposide in patients with advanced, refractory solid tumors and/or ES-SCLC. In addition, evaluate the toxicity and tolerability of AT-101 with cisplatin, etoposide, and Neulasta.

III. To evaluate the antitumor activity of this combination per tumor measurements using the Response Evaluation Criteria In Solid Tumors (RECIST) criteria.

SECONDARY OBJECTIVES:

I. To evaluate the pharmacokinetics of AT-101 as a single agent and in combination with cisplatin and etoposide in plasma.

II. To perform pharmacodynamic studies (genotyping of drug metabolizing enzymes, gene expression, and proteomics of drug-related pathways) on archived blood samples from patients treated with AT-101 in combination with cisplatin and etoposide.

OUTLINE: This is a dose-escalation study of R-(-)-gossypol.

Patients receive oral R-(-)-gossypol twice daily on days 1-3, cisplatin intravenously (IV) over 60 minutes on day 1*, and etoposide IV over 30 minutes on days 1*-3. Treatment repeats every 21 days for up to 6 courses during the dose escalation and 4 courses in the expanded extensive stage small cell lung cancer cohort, in the absence of disease progression or unacceptable toxicity.

Blood samples are collected on day 1 of courses 1 and 2 for pharmacokinetic analysis, biomarker assays, and correlative studies.

After completion of study treatment, patients are followed for 30 days.

[Note: *Cisplatin and etoposide will be started on day 2 during course 1; they will be given on day 1 during all subsequent courses.]

ELIGIBILITY:
Inclusion Criteria:

* In the dose-escalation cohorts: patients must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective; in the MTD expansion cohort: patients must have histologically or cytologically confirmed extensive-stage small cell lung cancer
* Patients must not have received prior therapy that inhibits the B-cell lymphoma 2 (Bcl-2) family
* Patients with small cell lung cancer may have received prior prophylactic cranial irradiation
* Prior whole brain radiotherapy allowed for patients with brain metastases provided they have stable/improved lesions for at least 1 month following treatment, no neurological symptoms and not require corticosteroids; an magnetic resonance imaging (MRI) of the brain or computed tomography (CT) scan of the head must be performed at baseline if patient has a history of brain metastases
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 12 weeks
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin < 1.5 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Serum creatinine < 1.5 x institutional upper limit of normal OR
* Creatinine clearance >= 45 mL/min/1.73 m^2, as calculated by Cockroft-Gault formula, for patients with creatinine levels above institutional normal; a 24 hour urine collection and creatinine clearance can be measured if indicated
* The effects of AT-101 on the developing human fetus are unknown; for this reason and because other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for at least one month following the last dose of AT-101; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients should display the ability to understand and the willingness to sign a written informed consent document
* Female patients of child bearing potential must not be pregnant
* Patients must have measurable or evaluable disease

Exclusion Criteria:

* Patients without small cell lung cancer who have had chemotherapy, radiotherapy or hormonal therapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered (=< grade 1) from clinically significant adverse events due to agents administered more than 4 weeks earlier; prior treatment with a platinum-based chemotherapy regimen in combination with thoracic radiation therapy is allowed for patients with ES-SCLC provided that recurrence of the SCLC occurred more than 6 months from definitive therapy for limited-stage small cell lung cancer; no other prior chemotherapy is allowed for the patients with ES-SCLC
* Failure to recover fully (as judged by the investigator) from prior surgical procedures
* Concurrent treatment with an investigational agent other than the investigational agent(s) used in this study OR treatment within 4 weeks of study entry with any investigational agent(s) or device(s)
* Any prior use of racemic gossypol or AT-101
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AT-101 or other agents used in study
* Requirement for routine use of hematopoietic growth factors (including granulocyte colony stimulating factor, granulocyte macrophage colony stimulating factor, or interleukin-11) or platelet transfusions to maintain absolute neutrophil counts or platelets counts above the required thresholds for study entry; if patient requires routine use of erythropoietin, eligibility at investigator discretion
* Any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain AT-101 tablets
* Patients with malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel are excluded; subjects with ulcerative colitis, inflammatory bowel disease, or a partial or complete small bowel obstruction are also excluded
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because the effects of AT-101 on the developing human fetus are unknown, but could potentially include teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AT-101, breastfeeding should be discontinued if the mother is treated with AT-101; these potential risks may also apply to other agents used in this study
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with AT-101 or other agents used in this study; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Patients with > grade 2 symptomatic hypercalcemia (based on investigator discretion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-09; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Toxicity and tolerability of R-(-)-gossypol acetic acid in combination with cisplatin and etoposide in terms of types and severities by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | Assessed up to 30 days after completion of study treatment
  The 95% confidence interval will be obtained.
Response as assessed by RECIST criteria | Assessed up to 30 days after completion of study treatment
  Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease. A 95% confidence interval of the overall response rate will be constructed.

SECONDARY OUTCOMES:
Pharmacokinetics of R-(-)-gossypol acetic acid in combination with cisplatin and etoposide | Days 1 and 2 of courses 1 and 2
  Summarized by dose level with simple summary statistics: means, medians, ranges, and standard deviations.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Traynor, Principal Investigator — University of Wisconsin, Madison
Locations (4):
- United States (4):
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Gundersen Lutheran, La Crosse, Wisconsin
  - UW Health Oncology - 1 South Park, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin